CLINICAL TRIAL: NCT02950688
Title: Evaluation of Correlates of Protective Efficacy of Seasonal Live Attenuated Influenza Vaccine (LAIV) by Utilization of a Human Challenge Model of Infection With Wild-type (wt) Influenza A/California/2009 (H1N1)-Like Virus
Brief Title: Safety and Effectiveness of a Seasonal Live Attenuated Influenza Vaccine in a Human Challenge Model of Infection With Wild-type (wt) Influenza A/California/2009 (H1N1)-Like Virus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: URMC 15-001
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Seasonal LAIV (Experimental): Participants will receive 1 dose of seasonal LAIV on Day 0. They will receive 1 dose of the wild-type A/California/2009-like influenza challenge virus on Day 56.
  Interventions: Biological: Seasonal LAIV; Biological: Wild-type A/California/2009-like Influenza Virus
- Group 2: Placebo (Placebo Comparator): Participants will receive 1 dose of placebo on Day 0. They will receive 1 dose of the wild-type A/California/2009-like influenza challenge virus on Day 56.
  Interventions: Biological: Placebo; Biological: Wild-type A/California/2009-like Influenza Virus

INTERVENTIONS:
Biological: Seasonal LAIV — 10^7.0 fluorescent focus units (FFU); administered by intranasal spray
  Other Names: FluMist Quadrivalent®
  Arms: Group 1: Seasonal LAIV
Biological: Placebo — Administered by intranasal spray
  Arms: Group 2: Placebo
Biological: Wild-type A/California/2009-like Influenza Virus — Approximately 3.5 x 10^6 TCID50; administered intranasally

SUMMARY:
The purpose of this study is to evaluate the immune response produced by a seasonal live attenuated influenza vaccine (LAIV) when compared to placebo. The initial vaccination will be followed 2 months later by an inpatient trial evaluating safety, infectivity, clinical response, and viral shedding after exposure to the wild-type A/California/2009-like influenza challenge virus.

DETAILED DESCRIPTION:
This study will evaluate the immune response produced by a seasonal LAIV. The initial vaccination will be followed 2 months later by an open-label inpatient trial evaluating the subsequent response (safety, infectivity, clinical response, and viral shedding) following administration of the wild-type A/California/2009-like influenza challenge virus.

Healthy adult participants will be randomized into two groups. On Day 0, Group 1 will receive a single dose of an intranasal LAIV. Group 2 will receive a single dose of intranasal placebo. Study visits will occur on Days 0, 3, 7, 14, and 28.

On Day 54, participants will be admitted to the isolation unit for the inpatient portion of the study, and both groups will receive an intranasal dose of wild-type A/California/2009-like influenza challenge virus on Day 56. On Day 65, participants who are no longer shedding virus will be discharged.

Follow-up study visits will occur after discharge from the isolation unit on Days 70, 84, 112, and 180. Study visits during either the inpatient or outpatient portions of the trial may include physical examinations, collection of blood and urine samples, electrocardiogram (ECG), nasal washes and swabs, and nasal mucus weighing.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 years and 45 years of age. Children will not be recruited or enrolled in this study for safety considerations and because of the need for isolation.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
* Likely to be susceptible to the challenge virus as determined by a baseline serum HAI antibody titer to the A/California/09 wild-type virus of 1:8 or less.
* Agree to storage of blood specimens for future research.
* Available for the duration of the trial.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Female subjects must agree to use effective birth control methods for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse, surgical sterilization). All female subjects will be considered being of child-bearing potential except those who have undergone hysterectomy and those in whom menopause occurred at least 1 year prior to the study.

Exclusion Criteria:

* Pregnancy as determined by a positive human choriogonadotropin (beta-HCG) test.
* Currently breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, endocrinologic or renal disease by history, physical examination, and/or laboratory studies including urine testing. Levels of alanine aminotransferase (ALT), aspartate transaminase (AST), bilirubin greater than 2 times the upper limit of normal (ULN) or otherwise clinically significant as determined by the Principal Investigator (PI), will be exclusionary at baseline, prior to vaccination. Complete blood count (CBC) with differential outside of the normal reference range and deemed clinically significant by the PI.
* Body Mass Index (BMI) of less than 18.5 or greater than 40.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* History of anaphylaxis.
* Allergy to oseltamivir as determined by subject report.
* Current diagnosis of asthma or reactive airway disease (within the past 2 years).
* History of Guillain-Barré Syndrome.
* Known immunodeficiency syndrome.
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination.
* Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) or any unlicensed vaccine within 6 months of enrollment.
* History of a surgical splenectomy.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Current smoker unwilling to stop smoking for the In-patient Challenge Phase of the study.

  * A current smoker includes anyone stating they currently smoke any amount of a tobacco product.
  * The decision to exclude a potential subject is determined by medical history and a clinician's clinical judgment based on the physical examination.
  * After admission to the unit, nicotine patches will be provided to current smokers who request them for the inpatient portion of the study.
* Allergy to eggs or egg products.
* Household contacts of individuals at higher risk for influenza-related complications, including: Persons greater than or equal to 65 years of age or less than 5 years of age; or persons with chronic pulmonary disease (e.g., asthma, emphysema), chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, ischemic heart disease), metabolic disease (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies), immunosuppression, neurological and neurodevelopmental conditions, children and teenagers who are receiving long-term aspirin therapy, or women who are pregnant or who are trying to become pregnant.
* Positive urine drug toxicology test indicating narcotic use/dependency.
* Positive ELISA and confirmatory tests for human immunodeficiency virus-1 (HIV-1), hepatitis C virus (HCV), or hepatitis B (Positive hepatitis B virus surface antigen).
* Clinically significant abnormalities on ECG.
* Clinically significant abnormality as deemed by the PI on echocardiographic testing.
* Known close contact with anyone known to have influenza or influenza-like illness in the past 7 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of any reactogenicity events after administration of seasonal LAIV | Measured through Day 180
Frequency of significant increases in nasal secretion hemagglutination (HA)-specific antibody assessed by enzyme-linked immunosorbent assay (ELISA) | Measured through Day 84
Frequency of instances of greater than 200 influenza-specific interferon-gamma-secreting cells per million lymphocytes as assessed by enzyme-linked immuno spot assay (ELISPOT) | Measured on Day 28 after immunization
Frequency of detection of influenza-specific immunoglobulin G (IgG) or immunoglobulin A (IgA) secreting B cells assessed by antibody secreting cells (ASC) assay | Measured on Day 7 following vaccination
Frequency of challenge virus shedding on one or more days on Days 56-63 as assessed by culture or real-time reverse transcriptase polymerase chain reaction (rRT-PCR) | Measured through Day 63
A 4-fold or greater increase in either hemagglutination-inhibition (HAI) or microneutralization (MN) antibody when compared to pre-challenge samples, as assessed by HAI assays | Measured through Day 56
A 4-fold or greater increase in either hemagglutination-inhibition (HAI) or microneutralization (MN) antibody when compared to pre-challenge samples, as assessed by MN assays | Measured through Day 56
A 4-fold or greater increase in either hemagglutination-inhibition (HAI) or microneutralization (MN) antibody when compared to pre-challenge samples, as assessed by blood serum titer | Measured through Day 56
Clinical symptoms recording of 10 key influenza symptoms (cough, sore throat, stuffy nose, dyspnea, fatigue, headache, myalgias, nausea, diarrhea, and feverishness) on an analog scale of severity | Measured through Day 180
Area under the curve (AUC) of symptom severity | Measured through Day 180
Total nasal mucus weight | Measured through Day 180
  Nasal mucus weights will be determined by collecting tissues over 24 hours, weighing them and subtracting the dry weight.

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States